CLINICAL TRIAL: NCT06729528
Title: Diagnostic Value of PePCI and ManTIS Scores in Whole-Body Computed Tomography (WBCT) Decision-Making for Pediatric Trauma Patients in the Emergency Department
Brief Title: Diagnostic Value of Whole-Body Computed Tomography (WBCT) Scores in Pediatric Trauma Patients
Status: Completed | Type: Observational
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emre Kudu, Assistant Professor, Marmara University Pendik Training and Research Hospital
Other Study IDs: 09.2024.782
Record Dates: First submitted 2024-11-27; First posted 2024-12-11 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Whole Body Computed Tomography Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Traumatic pediatric patients: Patients under 18 years old present to the emergency department red area due to trauma.
  Interventions: Diagnostic Test: The PePCI and ManTIS scores

INTERVENTIONS:
Diagnostic Test: The PePCI and ManTIS scores — The PePCI and ManTIS scores have been developed to predict the indication for whole-body CT in pediatric cases presenting to the emergency department with trauma. These scores help reduce unnecessary radiation exposure in pediatric trauma cases.

SUMMARY:
Pediatric trauma assessment is challenging due to difficulties in obtaining information, which increases the need for unnecessary imaging. Trauma-related injuries remain a significant cause of death in children. Although whole-body computed tomography (CT) is frequently used due to a lower threshold for imaging, issues such as high radiation exposure arise.

To reduce unnecessary radiation exposure in pediatric trauma patients, scoring systems such as PePCI (Pediatric Polytrauma CT Indication Score) and ManTIS (Manchester Trauma Imaging Score) have been developed. These studies have demonstrated their effectiveness in predicting the need for CT scans and preventing unnecessary examinations. However, both studies are retrospective analyses limited to a single region. Therefore, a prospective study is planned in Türkiye to evaluate the reliability and applicability of these scoring systems and their real-world benefits.

DETAILED DESCRIPTION:
The assessment of trauma in children is challenging due to difficulties in obtaining information about the mechanism and process of trauma, which leads doctors to perform more imaging. Although the incidence of fatal injuries in children has decreased in the last decade, trauma-related injuries remain a leading cause of death among children over one-year-old. Due to the lower imaging threshold in children compared to adults, whole-body computed tomography (WBCT) is frequently used. WBCT is an essential tool for the rapid diagnosis of injuries, especially in hemodynamically unstable pediatric multi-trauma patients.

The most accurate criteria for activating the trauma team in pediatric trauma patients are still being debated. According to the Advanced Trauma Life Support (ATLS) guidelines, the trauma team is activated based on the mechanism of injury; thus, WBCT is performed even in hemodynamically stable pediatric patients. This situation leads to unnecessary radiation exposure, increased costs, and resource wastage. Although the mechanism of injury does not constitute a sufficient indication for WBCT in pediatric patients, many trauma patients are evaluated with WBCT to avoid missing potential injuries.

In pediatric emergency department patients, it is known that WBCT is not associated with a reduction in mortality but is linked to high radiation exposure and increased lifetime risk for leukemia, solid cancers, and brain tumors. Therefore, although we know the benefits of targeted emergency CT scans, the usefulness of WBCT imaging for pediatric trauma patients is debated.

The severity of injuries, especially in multi-trauma patients, is classified using the Injury Severity Score (ISS). The ISS is based on an anatomical ordinal scale ranging from 1 to 75 points, with low scores representing mild injuries and high scores representing severe and fatal injuries. Generally, an ISS >15 indicates serious injuries. This scoring system is also applicable to children and adolescents. However, pediatric patients show lower mortality for the same ISS compared to adults, attributed to physiological response differences between adults and children. Therefore, a new classification for injury severity in pediatric patients has been proposed. While an ISS >15 in adults indicates serious injury, an ISS >23 in the pediatric population indicates serious injury, and patients with an ISS >26 may have functional impairments at discharge.

To reduce unnecessary radiation exposure and prevent resource wastage in pediatric trauma patients, a new study was conducted by Strahl and colleagues. The study involved pediatric emergency patients with high-energy trauma mechanisms at a Level I trauma center in Germany. As a result of this study, a pediatric polytrauma CT indication score (PePCI) was developed to analyze pediatric trauma patients and reduce radiation exposure. The performance of this score was compared with the ISS. In this study, cases were screened retrospectively. It was found that WBCT was applied to 243 pediatric trauma patients. If the PePCI score had been applied to pediatric trauma patients, it could have been determined that WBCT would not have been necessary for 76 of the 243 patients they screened. Moreover, no significant injuries would have been overlooked.

Another single-center study conducted by Davies and colleagues in the United Kingdom (UK) demonstrated that a large patient group in the UK is exposed to unnecessary radiation. This situation is thought to increase the risk of life-threatening outcomes, such as malignancy, in the future. With appropriate evaluation, it has been shown that WBCT imaging may not be necessary for some trauma patients. A scoring system called the Manchester Trauma Imaging Score (ManTIS) has been developed to facilitate this evaluation. The ManTIS score has been shown to safely reduce the number of unnecessary WBCTs in the young patient group.

Although these studies have shown that the PePCI and ManTIS scores effectively predict the need for WBCT and prevent unnecessary scans, they have been conducted in a single region. The developed scoring systems are only applicable to specific geographical areas. Additionally, both studies were retrospective. Therefore, this study plans to prospectively evaluate the reliability, applicability, and practicality of these scores in clinical practice in Türkiye, assessing their real-life benefits.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric trauma patients who present to the emergency red zone or are deemed appropriate for monitoring in the red zone during their emergency department visit.
* Patients for whom consent to participate in the study is provided by their legal guardians (as children are not able to provide consent independently)

Exclusion Criteria:

* Patients who have previously been included in the study.
* Patients who refuse treatment before their assessment is completed or withdraw their consent to participate in the study.
* Patients with incomplete study data.
* Patients with penetrating injuries

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes all pediatric trauma cases that present to the red area of the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Whole Body Computed Tomography Need | through study completion, an average of 8 months
  Patients will be evaluated by an expert panel, which will include three emergency medicine specialists. The panel will assess all relevant clinical data, including trauma history, physical examination findings, laboratory results, imaging outcomes, consultations, and final dispositions. Based on this comprehensive evaluation, the panel will determine whether the patient requires WBCT. As a result, the primary outcome will be recorded as a binary measure: either the patient requires WBCT or does not require WBCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strahl A, Willemsen JF, Schoof B, Reinshagen K, Frosch KH, Wintges K. The paediatric polytrauma CT-indication (PePCI)-score-Development of a prognostic model to reduce unnecessary CT scans in paediatric trauma patients. Injury. 2024 May;55(5):111494. doi: 10.1016/j.injury.2024.111494. Epub 2024 Mar 11. PMID 38521635
- [Background] Davies RM, Scrimshire AB, Sweetman L, Anderton MJ, Holt EM. A decision tool for whole-body CT in major trauma that safely reduces unnecessary scanning and associated radiation risks: An initial exploratory analysis. Injury. 2016 Jan;47(1):43-9. doi: 10.1016/j.injury.2015.08.036. Epub 2015 Sep 1. PMID 26377772